CLINICAL TRIAL: NCT00598182
Title: From Immediate-release MPH to OROS MPH: The Impact Upon Family of Children and Adolescents With ADHD
Brief Title: Adherence and Long-term Effect of OROS Methylphenidate (CONCERTA): A Follow-up Study
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200709022R
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Disorder with Hyperactivity; OROS methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objectives of this study are to investigate:

1. the evolution of ADHD symptoms, remission rate of ADHD, social and school function, and familial relationship;
2. the adherence to CONCERTA, treatment modality, and average treatment duration during the 3-year follow-up period; and
3. the effect of medication on the changes of neuropsychological functioning.

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is a common impairing disease among children and adolescents. Methylphenidate, a stimulant, is effective in treating these patients. OROS methylphenidate (CONCERTA) provides ADHD patients a more convenient and safer treatment approach than immediate-release methylphenidate (IR-MPH). However, there is little information of long-term effect and adherence to CONCERTA. At the NTUH Taiwan, a randomized clinical trial of OROS MPH was performed 3 years ago and 64 subjects were included and treated with either IR MPH or OROS MPH followed by OROS MPH. Therefore, we purpose this study to follow up these patients, exploring the adherence rate to CONCERTA, symptoms evolution, and outcomes among these patients.

Overview of Study Design: There will be two stages of this study. All study procedures will be performed after obtaining informed consent.

Stage I: Medical charts of these subjects will be reviewed to obtain information about CONCERTA adherence (also including dosage, treatment duration, clinic visits, missing visits etc.), psychiatric co-morbidities, and other treatment approaches subjects received after the previous study. Subjects will be visited (Visit 1) and the information of baseline characteristics and reasons for discontinuing CONCERTA (if applicable) will be recorded. The assessments will included parent or teacher ratings on the Conner's Teacher and Parent Rating scales (CPRS-R:S, CTRS-R:S), the SNAP-IV rating scale, the SKAMP rating scale, investigator ratings on the Kiddie-SADS-E, Clinical Global Impression and the Social Adjustment Inventory for Children and Adolescents (SAICA); and neuropsychological assessments (Conner's Continuous Performance Test, CPT, and Cambridge Neuropsychological Test Automated Batteries, CANTA B) will be performed to these subjects.

Stage II: All subjects enrolled into stage one will be followed for the next 6 months. Medication for ADHD treatment may be used to these subjects based on investigators' clinical judgments. Subjects will visit clinics in week-24 (Visit 2). The same assessments at Visit 1 will be performed at Visit 2. In addition, the adherence to treatment, adverse events, overall satisfaction to treatment, and academic performances during these 6 months will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated the randomized clinical trial for CONCERTA on NTUH.
* Subjects whose parents/caregivers can complete the questionnaires during the study and can assist to finish the assessment properly during the study;
* Subjects whose parent(s) or guardian(s) has signed and dated an informed consent for the subject to participate in the study.

Exclusion Criteria:

* No.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who were diagnosed as DSM-IV ADHD and participated in the randomized clinical trial for CONCERTA at NTUH Taiwan will be enrolled into this study.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2007-09; Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan